CLINICAL TRIAL: NCT02852369
Title: Task Oriented Training and Evaluation at Home (TOTE Home)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowe, Veronica, M.D. (Individual)
Responsible Party: Principal Investigator, Veronica Rowe, Doctoral Student, Rowe, Veronica, M.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOTE Home 001
Record Dates: First submitted 2016-07-27; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Task Oriented Training (Experimental): The intervention administered during each of the training sessions was modeled after the protocol outlined in Winstein et al. (2013) however implementation was in the participant's home setting and involved tasks in the participant's real world.
  The manual entitled, "Upper-Extremity Task-Specific Training After Stroke or Disability" by Lang and Birkenmeier (2014) was also utilized to give a general overview of task specific training for the upper extremity and to help guide each activity the participant chose to work on.
  Interventions: Behavioral: Task Oriented Treatment

INTERVENTIONS:
Behavioral: Task Oriented Treatment — The intervention administered during each of the training sessions was modeled after the protocol outlined in Winstein et al. (2013) however implementation was in the participant's home setting and involved tasks in the participant's real world.
  The manual entitled, "Upper-Extremity Task-Specific Training After Stroke or Disability" by Lang and Birkenmeier (2014) was also utilized to give a general overview of task specific training for the upper extremity and to help guide each activity the participant chose to work on.

SUMMARY:
Objective: To determine the effectiveness of an upper extremity, task oriented training program delivered at home (TOTE Home) for people who are in the subacute recovery phase of a stroke.

Method: A single-subject AB series design with a follow-up to assess the effectiveness of TOTE Home which includes a maximum of 30, one hour sessions of training conducted in participants' homes. Repeated target measures of accelerometry and level of confidence to be analyzed throughout the study. Change scores from standardized assessments to be evaluated at baseline, post-intervention, and follow-up time periods.

DETAILED DESCRIPTION:
Hemiparesis following a stroke frequently leads to "learned non-use" of the weaker arm and hand. Task oriented training has been suggested as a contemporary neurorehabilitation technique. A single-subject AB series design with a follow-up was conducted to assess the effectiveness of a task oriented training program administered in participants' homes. This intervention, Task Oriented Training at Home (TOTE Home), incorporated current experience-dependent plasticity aspects modeled after the Acquired Skill Acquisition Program (ASAP) protocol parameters and principles of task oriented training as suggested by Lang and Birkenmeier in 2014. Repeated measures of accelerometry and level of confidence on a priority task were analyzed with visual analysis of changes in level, trend, and slope. Change scores from standardized assessments for the upper extremity, Motor Activity Log, Stroke Impact Scale question of recovery, Functional Test for the Hemiparetic Upper Extremity, and Canadian Occupational Performance Measure were evaluated on data collected at baseline, post-intervention, and follow-up time periods.

ELIGIBILITY:
Inclusion Criteria:

* upper extremity hemiparesis due to a stroke but met minimal movement criteria in the affected arm and hand (at least 10 degrees of active movement at the wrist, elbow, and shoulder movement, along with 10 degrees of active movement in the thumb and two other fingers)
* minimal cognitive deficits as demonstrated by a 24 or higher on the Mini-Mental Status Exam
* able to identify at least five specific tasks participants wish to achieve with their affected upper extremity. This was assessed with the Canadian Occupational Performance Measure (COPM)
* at least 21 years of age
* able to communicate in English
* 3-12 months after their stroke which would classify them in the subacute level of recovery
* all formal occupational therapy was completed.

Exclusion Criteria:

* upper extremity pain that interfered with activities of daily living
* requiring maximal assistance for mobility
* arm or hand injury (unrelated to the stroke)
* upper extremity amputations
* inability to participate due to any illness, social or geographical reason, and any other diagnosis or limiting conditions that would affect participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Movement of the hemiparetic upper extremity as measured by accelerometry | 24 hour recordings over 8 day periods

CONTACTS AND LOCATIONS:
Overall Officials: Marsha Neville, PhD, OT, Study Chair — Texas Woman's University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rowe VT, Neville M. Task Oriented Training and Evaluation at Home. OTJR (Thorofare N J). 2018 Jan;38(1):46-55. doi: 10.1177/1539449217727120. Epub 2017 Aug 31. PMID 28856960